CLINICAL TRIAL: NCT06714916
Title: Mutimodal Artificial Intelligence for Optimising Renal Tumour Management: Diagnosis, Surgery and Prognosis
Brief Title: Optimising Renal Tumour Management Through Artificial Intelligence Modules
Status: Recruiting | Type: Observational
Sponsor: Shao Pengfei (Other)
Responsible Party: Sponsor-Investigator, Shao Pengfei, chief physician, The First Affiliated Hospital with Nanjing Medical University
Organization: The First Affiliated Hospital with Nanjing Medical University (Other)
Other Study IDs: 2024-SR-961
Record Dates: First submitted 2024-12-02; First posted 2024-12-04 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2024-12

CONDITIONS: Renal Neoplasms; Pathology; Renal Cell Cancer
Keywords: Articicial Intelligence; Renal tumors; Prediction Model; Surgery; Radiomics; Pathomics
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to improve the management of people with renal tumour by multimodal artificial intelligence(AI). It will also measure the accuracy of the predictions from AI models. The main questions it aims to answer are:

1. whether the AI module can accurately provide tumor-related information such as Benign or malignant, subtypes, grading, stage, etc. by learning from preoperative CT images.
2. whether the AI module can help clinicians find out the most suitable surgical programme for people with renal tumor.
3. whether the AI module can integrate CT images and pathology slides, offering supplementary prognostic information to improve postoperative survival.

Participants who complete a CT(usually Contrast-enhanced CT, CECT) examination and undergo radical or partial nephrectomy will carry out active surveillance and record postoperative survival data for 5 years.

DETAILED DESCRIPTION:
In this study, AI model will explore and clarify features in renal tumor CT images and pathological images that are difficult to detect manually, and then correlate them with clinical outcomes, thereby improving the diagnosis and treatment process for renal tumors. Firstly, the model can accurately distinguish renal tumor subtypes and predict stage, grade, and complexity so as to svoid misdiagnosis and assist clinicians in formulating treatment plans. Secondly, by learning from surgical videos, the model can provide additional information during surgerys, such as important anatomical landmarks, location of tumors. Finally, combining radiomics and pathomics, the model can differentiate between high-risk and low-risk patients after surgery, thus providing personalized prognostic guidance.

ELIGIBILITY:
Inclusion Criteria:

* Patients with renal tumor which can be treated by surgery;
* Complete CECT within 30 days before surgery;
* Patients who fully understand this study and sign the informed consent;

Exclusion Criteria:

* Patients with any item missing from the baseline clinical and pathological information;
* Patients who has already metastasized by the time the tumor is discovered;
* Previous treatment in any form, including surgery, targeted therapy and immunotherapy;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with renal tumors on imaging examinations who underwent surgery
Sampling Method: Non-Probability Sample
Enrollment: 2100 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessing the performance of AI models by the "AUC" comprehensive assessment model | From enrollment to the end of 5-years' follow up
  "AUC" refers to the area under the ROC (Receiver Operating Characteristic) curve, which indicates the performance of the model in predicting immunohistochemistry-related pathological information of prostate cancer after surgery, and the AUC ranges from 0-1, with the larger value indicating the better prediction effect.

SECONDARY OUTCOMES:
Assessing the model's performance to predict participants' prognosis post-surgery by Kaplan-Meier Survival Analysis | From enrollment to the end of 5-years' follow up
  Kaplan-Meier Survival Analysis s a non-parametric statistic mainly used to figure out factors which indicate survival.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University (Jiangsu Provincial People's Hospital), Nanjing, Jiangsu, China